CLINICAL TRIAL: NCT06092892
Title: IIT2023-09-Chung-UpfrontTAD: Upfront TAD/SNB in Patients With Clinical T1-2N0 ER+ Her2- Breast Cancer With Ultrasound Detected Nodal Metastases
Brief Title: IIT2023-09-Chung-UpfrontTAD: Upfront TAD/SNB in Patients With Breast Cancer With Nodal Metastases
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Alice Chung (Other)
Responsible Party: Sponsor-Investigator, Alice Chung, Sponsor-Investigator, Cedars-Sinai Medical Center
Organization: Cedars-Sinai Medical Center (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IIT2023-09-Chung-UpfrontTAD
Record Dates: First submitted 2023-10-16; First posted 2023-10-23 (Actual); Last update posted 2025-12-10 (Actual); Status verified 2025-12

CONDITIONS: Breast Cancer; Axillary Nodal Disease; Female Breast Cancer; Axilla; Breast; Mastectomy; Lymphedema; Tumor, Breast
Keywords: T1-2N0 ER+ invasive; biopsy; upfront lumpectomy
MeSH Terms: conditions — Breast Neoplasms; Lymphedema | interventions — Mastectomy, Segmental; Mastectomy

STUDY DESIGN:
Intervention Model Description: Open label, single arm
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Single Arm (Experimental)
  Interventions: Procedure: Breast Surgery (BCS or mastectomy) with TAD/SNB; Radiation: Adjuvant Radiation Therapy

INTERVENTIONS:
Procedure: Breast Surgery (BCS or mastectomy) with TAD/SNB — Breast surgery (BCS or mastectomy) with TAD/SNB & Adjuvant Radiation therapy
Radiation: Adjuvant Radiation Therapy — Breast surgery (BCS or mastectomy) with TAD/SNB & Adjuvant Radiation therapy

SUMMARY:
The purpose of the study is to determine the recurrence rates and survival of patients with clinical T1-2N0 ER+/Her2- invasive breast cancer who have biopsy proven image detected nodal disease treated with upfront lumpectomy or mastectomy with TAD followed by adjuvant therapy. This is a prospective, single arm phase II clinical trial. Patients will be screened and enrolled per eligibility criteria. Patient, tumor, and treatment data will be documented.

ELIGIBILITY:
Inclusion Criteria:

* Women age ≥ 45
* Clinical T1-2N0 ER+ invasive breast cancer
* US detected biopsy proven axillary nodal disease
* Written informed consent obtained from subject and ability for subject to comply with the requirements of the study.

Exclusion Criteria:

* Palpable nodes on physical exam
* Her2+ or ER- invasive breast cancer
* Extranodal extension > 3 mm on nodal biopsy
* More than 2 suspicious nodes on preoperative imaging

Min Age: 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Estimated)
Dates: Start 2024-04-07 (Actual); Primary Completion 2031-04 (Estimated); Study Completion 2031-04 (Estimated)

PRIMARY OUTCOMES:
Regional recurrence rate | 5 Years
  Regional recurrence rate is defined as the percentage of patients who experience a regional recurrence during follow-up period.

SECONDARY OUTCOMES:
Local recurrence rate | 5 Years
  Local recurrence rate is defined as the percentage of subjects who experience a local recurrence during follow-up period.
Disease-free survival (DFS) | 5 Years
  Disease-free survival (DFS) is defined as the length of time after targeted axillary dissection (TAD) that the subject survives without any signs or symptoms of breast cancer.
Breast cancer specific survival (BCSS) rate | 5 Years
  Breast cancer specific survival (BCSS) rate is defined as the percentage of subjects who have not died from breast cancer during follow-up period
Overall survival (OS) | 5 Years
  Overall survival (OS) is defined as the length of time from targeted axillary dissection (TAD) that the subjects are still alive.

CONTACTS AND LOCATIONS:
Overall Officials: Alice Chung, MD, Principal Investigator — Cedars-Sinai Medical Center
Locations (3):
- United States (3):
  - Cedars-Sinai Medical Center, Samuel Oschin Comprehensive Cancer Institute, Los Angeles, California
  - CS Cancer at Huntington Cancer Center, Pasadena, California
  - CS Cancer at Valley Oncology Medical Group, Tarzana, California

IPD SHARING:
Plan to Share IPD: No